CLINICAL TRIAL: NCT05168514
Title: The Effect of Back Massage on Palliative Care Patients on Sleep Quality and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Sevil PAMUK CEBECİ, Asst.Prof.Dr., Eskisehir Osmangazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-2
Record Dates: First submitted 2021-12-09; First posted 2021-12-23 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Palliative Care
Keywords: back massage; Palliative care; nursing care; massage practice; pain; sleep quality
MeSH Terms: conditions — Pain; Sleep Initiation and Maintenance Disorders | interventions — Massage

STUDY DESIGN:
Masking Description: Single-blind randomized control method will be used in the study, patients in the experimental and control groups will not know which group they are in. Randomization Method: Experimental and control groups will be determined from patients who meet the sampling selection criteria, using the Random Integer Generator method from the random.org site, Numbersalt.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Massage (Experimental): Massage begins with the patting (eflorage) maneuver. Massage is continued with petrissage, bearing, friction and percussion maneuvers.
  Maneuvers are performed for 3-5 minutes. A patting motion is performed between maneuvers and at the end of the massage. During the massage, it is observed whether the integrity of the skin is impaired or in terms of redness.
  Interventions: Other: Massage

INTERVENTIONS:
Other: Massage — "Patient Identification Form", "Pittsburgh Sleep Quality Index" and "McGill Pain Scale Short Form" will be applied to patients with written and verbal consent. Scales and massage application will be done before the pharmacological agent is administered to the patients.
  Back massage will be applied to the experimental group for 10 minutes every day for 10 days. Routine treatment and care practices in the clinic will continue. "Pittsburgh Sleep Quality Index", "McGill Pain Scale Short Form" will be applied to the experimental group before and after each massage and scores will be recorded for 10 days.
  The control group will not be interfered with, and the routine treatment and care practices in the clinic will continue. "Pittsburgh Sleep Quality Index", "McGill Pain Scale Short Form" will be applied to the control group simultaneously with the experimental group and scores will be recorded for 10 days.

SUMMARY:
This study was planned to evaluate the effect of back massage applied to palliative care patients on sleep quality and pain.

DETAILED DESCRIPTION:
The most common complaint in palliative care patients is pain. Therefore, the quality of palliative care is demonstrated by the good management of patients' pain and suffering. In the treatment of pain, pharmacological and non-pharmacological treatments should be used together. As a result of the relaxation of the muscles with massage, which is one of the non-pharmacological treatments, the pain is relieved and reduced. Again, massage increases the release of endorphins and reduces the feeling of pain. Another common complaint in palliative care patients is insomnia. Sleep quality is also linked to pain. Low sleep quality causes a decrease in tolerance to pain, more drugs are used to relieve pain, and a negative cycle is formed by affecting sleep quality. Massage is one of the oldest treatment methods used to relieve many ailments. Florence Nightingale described massage in her Notes on Nursing published in 1859 and provided its use in the field of nursing.

This study was planned to evaluate the effect of back massage applied to palliative care patients on sleep quality and pain.

The study was planned as a randomized controlled experimental study between November 2021 and June 2022. Patients hospitalized in the Palliative Care Service of Bilecik Training and Research Hospital, the sample will be 52 patients, 26 patients in each group, with a 95% CI 90% power, as a result of the calculation made using the G*Power 3.1.9.7 program. Written consent will be obtained from the patients who agree to participate in the study and the "Patient Identification Form" will be filled. Back massage will be applied to the experimental group for 10 minutes every day for 7 days. Pittsburgh Sleep Quality Index, McGill Pain Scale Short Form will be administered after each massage and scores will be recorded for 7 days. Scales and massage will be applied to the patients before the administration of the pharmacological agent, which is among the routine treatment and care practices in the clinic. The control group will not be interfered with, and the routine treatment and care practices in the clinic will continue. Pittsburgh Sleep Quality Index, McGill Pain Scale Short will be applied to the control group simultaneously with the experimental group and scores will be recorded for 7 days. The obtained data will be evaluated using appropriate statistical methods.

As a result of the research, it is thought that the questions of whether there is a significant difference in sleep quality and pain scale between the patient group who received back massage in palliative care and the patient group who did not receive it will be answered.

ELIGIBILITY:
Inclusion Criteria:

* At least literate education level,
* Having no cognitive, affective and verbal communication problems that would prevent the understanding of the given information and the ability to accurately express pain and sleep,
* Over 18 years old,
* Being in the palliative service,
* Patients who do not react negatively to any attempt to touch, such as massage,
* Patients with full and healthy tissue integrity in the area to be massaged.

Exclusion Criteria:

* İlliterate to read and write
* Having any cognitive, affective and verbal communication problems that prevent the understanding of the given information and the ability to accurately express pain and sleep,
* Under the age of 18,
* Reacts negatively to any attempt to touch, such as massage,
* Patients whose tissue integrity is not complete and healthy in the area to be massaged.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
To accept the hypothesis that there is a significant difference between the sleep quality mean scores of the experimental group and the sleep quality mean scores of the control group in palliative care patients. | 10 weeks
  The Pittsburgh Sleep Quality Index (PUKI) will be used to measure the effect of back massage applied to the experimental group on sleep quality. PUKI is a 19-item scale that evaluates sleep quality and disorder. Each item of the test is scored between 0-3. The scale consists of 7 subscales that assess subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disorders, use of sleep medication, and loss of daytime functionality. By summing up the subscales, a total PUKI score ranging from 0 to 21 is obtained. A total PSQI score greater than five, with 89.6% sensitivity and 86.5% specificity, indicates inadequate sleep quality and indicates severe impairment in at least two areas or moderate impairment in three areas.
To accept the hypothesis that "there is a significant difference between the mean pain score of the experimental group and the pain score of the control group in palliative care patients". | 10 weeks
  The scale consists of three parts; first part; 11 of them evaluate the sensory and 4 of them evaluate the perceptual dimension of the pain. These descriptors are rated on an intensity scale from 0 to 3 (0= none, 1= mild, 2= moderate, 3= excessive). In the first part of the scale, a total of three pain scores are obtained: sensory pain score, perceptual pain score and total pain score. The sensory pain score is between 0-33, the perceptual pain score is between 0-12, and the total pain score is between 0-45. The increase in the score indicates that the pain also increased. Part Two: There were five word groups ranging from "mild pain" to "unbearable pain" to determine the severity of the patient's pain. Part Three: The patient's current pain intensity was assessed using a visual comparison scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sevil PAMUK CEBECİ, Study Director — sevil.pamukcebeci@ogu.edu.tr
Locations (1):
- Bilecik Devlet Hastanesi, Bilecik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No